CLINICAL TRIAL: NCT00042328
Title: A Pharmacokinetic Study of Valacyclovir in Pediatric Oncology Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Susan Blaney, Professor, Baylor College of Medicine
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H9912; VALACYCLOVIR SINGLE DOSE
Record Dates: First submitted 2002-07-26; First posted 2002-08-01 (Estimated); Last update posted 2015-08-24 (Estimated); Status verified 2015-08

CONDITIONS: Neoplasms
Keywords: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Valacyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Valacyclovir

SUMMARY:
The purpose of this research is to study the pharmacology (how the body handles this drug) of valacyclovir in children receiving treatment for cancer. This study will last approximately 7 days.

DETAILED DESCRIPTION:
In this study, patients will receive a single dose of oral valacyclovir. Blood samples will be drawn to evaluate the pharmacology (how the body handles the drug). Blood samples (less than one teaspoon each) will be obtained before receiving the drug and at 0.5, 1, 1.5, 2, 5, 6, and 8 hours after receiving the drug. The total amount of blood drawn from patients for all blood work including routine blood tests as well as pharmacokinetics will not be greater than 5% of the total blood volume.

We will also have all urine output collected for 8 hours starting at the time patients receive the dose of valacyclovir. A 5cc sample of urine will be collected and analyzed to determine how the body handles the drug at hours 2, 4, 6, and 8.

ELIGIBILITY:
Inclusion criteria:

* Age: Patients must be > / = 2 and < / = 18 years old.
* Life Expectancy: Patients must have a life expectancy of > 8 weeks
* Subjects must have a diagnosed malignancy, and must currently be receiving consolidation or maintenance chemotherapy
* Hepatic/Renal Function: Patients must have adequate hepatic function (bilirubin < / = 1.5 mg/dl: SGPT < 3x normal) and adequate renal function (creatinine < / = 1 mg/dl: BUN < 20 )
* Medication Tolerance: Patients must be able to swallow pills or tolerate a suspension of the medication
* Fluid Tolerance: Children must be able to retain liquids at the time of enrollment
* Informed Consent: Written informed consent will be obtained from all patients and/or their parents prior to enrollment
* Pregnancy: Women of childbearing age must have a negative serum pregnancy test at the time of study entry

Exclusion criteria:

* More than one prior chemotherapy regimen.
* Patients with uncontrolled infections.
* Subjects with known history of adverse reaction to acyclovir in the past.
* Patients with concurrent infections requiring treatment with valacyclovir or acyclovir.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30
Dates: Start 2001-08; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Blaney, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States